CLINICAL TRIAL: NCT02366767
Title: Assessment of an Automatic Closed-loop Insulin Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce A. Buckingham, MD, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G140095
Record Dates: First submitted 2014-06-26; First posted 2015-02-19 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Insulin Infusion Systems; Continuous Glucose Monitors
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- automatic closed-loop insulin delivery (Experimental): The closed-loop arm will consist of participants wearing a sensor and transmitter which transmits sensor glucose data. The algorithm determines insulin delivery rates and this is delivered in microboluses every 5 minutes
  Interventions: Device: Automatic closed-loop insulin delivery
- Control (Active Comparator): The subjects in the control arm will wear the 530G system using Enlite and MiniLink transmitter and threshold suspend.
  Interventions: Device: Control

INTERVENTIONS:
Device: Automatic closed-loop insulin delivery — Sensor transmit glucose data every 5 minutes to the control algorithm which adjusts insulin delivery every 5 minutes.
  Arms: automatic closed-loop insulin delivery
Device: Control — Threshold suspend
  Other Names: 530G Pump
  Arms: Control

SUMMARY:
The overall aim of this research proposal is to determine the safety, feasibility and efficacy of an automatic closed-loop insulin delivery system.

DETAILED DESCRIPTION:
This study will be completed in two parts.

The initial part of this study will be an inpatient evaluation of the system with the primary goal of assessing safety and feasibility. This will involve 8 subjects with type 1 diabetes, aged 14 - 40 years, admitted for up to 60 hour. Plasma glucose levels will be collected hourly and tested by YSI (YSI 2300, Yellow Springs Instrument). These studies will be performed at Stanford University and will include group sporting activities to mimic the diabetes camp environment. Capillary blood glucose testing will be performed every 2-3 hours before meals, snacks, exercise, and prebed by subjects with research staff supervision during the day and at 00:00, 03:00 and 07:00 by research staff. These data will be reviewed by the DSMB before proceeding to camp studies.

The second part of this study will be to test the efficacy of the system during diabetes summer camps. We will test the system in subjects with type 1 diabetes, aged 14-40 years, attending diabetes camp. There will be 20 subjects recruited, with 10 subjects randomized to the control arm Medtronic 530G system with threshold suspend (control group) and 10 subjects randomized to the automatic closed-loop insulin delivery (intervention group). Capillary blood glucose testing will be performed every 2-3 hours before meals, snacks, exercise and prebed by subjects with research staff supervision and at 00:00, 03:00 and 07:00 by research staff. The primary aim of this study is to generate preliminary data of system safety and efficacy in a closely supervised environment that challenges glucose control.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes

   * The diagnosis of type 1 diabetes is based on the investigator's judgment
   * C peptide levels and antibody determinations are not required
2. Daily insulin therapy for ≥ 12 months
3. Insulin pump therapy for ≥ 3 months
4. Age 14.0 - 40.0 years
5. Subject comprehends written English
6. Female subjects who are sexually active must be on acceptable method of contraception e.g. oral contraceptive pill, diaphragm, IUD
7. Female subjects past menarche must have a negative urine pregnancy test
8. Informed consent form is signed by the subject and/or parent and assent assigned by the subject if under 18 years of age
9. For subjects under 18 years, both the subject and parent/guardian understand the study protocol and agree to comply with it. Both parents must sign if possible.

Exclusion Criteria:

1. Subject has a medical disorder that in the judgment of the investigator will affect the wearing of the devices or the completion of any aspect of the protocol
2. Diabetic ketoacidosis in the past month
3. Hypoglycemic seizure or loss of consciousness or an event requiring glucagon or IV glucose in the past 3 months
4. Subject has a respiratory condition such as asthma, treated with systemic or inhaled corticosteroids in the previous 6 months or cystic fibrosis
5. Subject has a history of any cardiac or vascular disorder such as myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, arrhythmia or thromboembolic disease
6. Subject has a history of liver or kidney disease (other than microalbuminuria)
7. Subject has active Graves' disease
8. Subjects with inadequately treated thyroid disease or celiac disease
9. Subject has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
10. Subject has a history of diagnosed medical eating disorder
11. Subject has a history of known illicit drug abuse
12. Subject has a history of known prescription drug abuse
13. Subject has a history of current alcohol abuse
14. Subject has a history of visual impairment which would not allow subject to participate
15. Subject has an active skin condition that would affect sensor placement
16. Subject has adhesive allergies
17. Subjects requiring an intermediate or long-acting insulin (such as NPH, detemir or glargine)
18. Subjects requiring other anti-diabetic medications other than insulin (oral or injectable)
19. Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
20. Subject is currently on beta blocker medication
21. Subject is currently participating in another investigational study (drug or device)
22. Subject is deemed by the investigator to be unwilling or unable to follow the protocol
23. Presence of a febrile illness within 24 hours of enrollment

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Camp Conrad-Chinnock, Angelus Oaks, California
  - Packard El Camino Hospital, Mountain View, California
  - Lucile Packard Children's Hospital, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ly TT, Roy A, Grosman B, Shin J, Campbell A, Monirabbasi S, Liang B, von Eyben R, Shanmugham S, Clinton P, Buckingham BA. Day and Night Closed-Loop Control Using the Integrated Medtronic Hybrid Closed-Loop System in Type 1 Diabetes at Diabetes Camp. Diabetes Care. 2015 Jul;38(7):1205-11. doi: 10.2337/dc14-3073. Epub 2015 Jun 6. PMID 26049550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for the Inpatients studies at Stanford were recruited from the Packard Diabetes clinics.
  Subjects for the camp studies were recruited from patients who had completed registration forms to attend camp. They were sent a letter describing the study and if they were interested they contacted us.
Pre-assignment Details: one subject enrolled in the closed-loop group had to leave camp after 24 hours and was replaced.
Period: Overall Study
Arm/Group | Automatic Closed-loop Insulin Delivery | Control
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — left for home after 1 day at camp | 1 | 0

BASELINE CHARACTERISTICS:
Population: type 1 diabetes attending a diabetes summer camp
Groups:
- Total: Total of all reporting groups
Arm/Group | Automatic Closed-loop Insulin Delivery | Control | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (4.7) | 17.7 (2.2) | 18.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 8.5 (1.9) | 8.6 (1.05) | 8.6 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Automatic Closed Loop Insulin Delivery System in Adolescents and Adults With Type 1 Diabetes
Description: 1. As measured by the number of events of plasma glucose values ≤ 50 mg/dL OR frequency of system alerts preceding a plasma glucose value of ≤ 50 mg/dL in all subjects
  2. As measured by the number of events of system alerts of plasma glucose values >300 mg/dL lasting for more than one hour in all subjects.
  3. As measured by number of events of serum ketones >3 mmol/L in all subjects
  4. As measured by the number of events meeting the criteria for severe hypoglycemia, defined as hypoglycemic seizure, loss of consciousness or coma or an event requiring administration of glucagon or IV glucose in all subjects
Time Frame: 6 days
Population: 10 subjects who completed study
Measure: Number; unit: Events
Arm/Group | Automatic Closed-loop Insulin Delivery | Control
Number analyzed (Participants) | 10 | 10
Events
  Plasma glucose <50 mg/dL | 9 | 6
  Plasma glucose >300 mg/dL lasting more than 1 hour | 0 | 0
  Serum Ketones >3 mmol/L | 0 | 0
  Severe Hypoglycemia | 0 | 1

2. Secondary Outcome: Feasibility of Using the Automatic Closed Loop Delivery System in Adolescents and Adults With Type 1 Diabetes
Description: 1. As measured by the system initiating and operating properly for at least 75% of the time for 75% of subjects.
  2. As measure by the completion of study enrollment procedures and education on system use within 2 hours for 75% of the subjects.
Time Frame: 6 days
Measure: Number; unit: participants
Arm/Group | Automatic Closed-loop Insulin Delivery | Control
Number analyzed (Participants) | 10 | 10
participants
  Operational System >75% time | 10 | 10
  Education completed within 2 hours | 10 | 10

3. Secondary Outcome: Efficacy of Hybrid Closed-loop System in Comparison With Control
Description: As measured by overall mean sensor glucose percent time in range 70-180 mg/dL.
Time Frame: 6 days
Population: Including only sensor data where the daily median ARD <15%.
Measure: Mean (Standard Error); unit: Percent time
Arm/Group | Automatic Closed-loop Insulin Delivery | Control
Number analyzed (Participants) | 10 | 10
Percent time | 69.9 (3.3) | 73.1 (5.0)

ADVERSE EVENTS:
Time Frame: 6 days of camp
Arm/Group | Automatic Closed-loop Insulin Delivery | Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Automatic Closed-loop Insulin Delivery (N=11) | Control (N=10)
hypoglcyemic seizure (Endocrine disorders) | 0 (0) | 1 (1) — Had seizure after taking dinner insulin and food was delayed

LIMITATIONS AND CAVEATS:
This study was in a closely supervised diabetes camp setting. There was close supervision of fingerstick testing using the second drop of blood. Research staff did not assist subjects in carbohydrate counting and meal sizes were unrestricted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No